CLINICAL TRIAL: NCT00473135
Title: Safety and Immunogenicity of a 2-Dose Regimen of rDEN1delta30 Dengue Serotype 1 Vaccine With Boosting at 4 Versus 6 Months
Brief Title: Safety of and Immune Response of a 2-dose Regimen of rDEN1delta30 Dengue Virus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Anna Durbin, MD, Center for Immunization Research, Johns Hopkins School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 229; WIRB Protocol Number 20070718
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2008-01

CONDITIONS: Dengue
Keywords: Dengue Fever; Dengue Vaccine; Dengue Virus; Dengue Hemorrhagic Fever; Dengue Shock Syndrome
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Two subcutaneous vaccinations with rDEN1delta30 into the deltoid region or either arm. One vaccination is given on Day 0 and one vaccination is given on Day 120.
  Interventions: Biological: rDEN1delta30
- 2 (Experimental): Two subcutaneous vaccinations with rDEN1delta30 into the deltoid region or either arm. One vaccination is given on Day 0 and one vaccination is given on Day 180.
  Interventions: Biological: rDEN1delta30
- 3 (Placebo Comparator): Two subcutaneous vaccinations with placebo into the deltoid region or either arm. One vaccination is given on Day 0 and one vaccination is given on either Day 120 or 180, depending on arm assignment.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: rDEN1delta30 — Live attenuated rDEN1delta30 vaccine at a dose of 10^3 PFU
  Arms: 1; 2
Biological: Placebo — Placebo for rDEN1delta30
  Arms: 3

SUMMARY:
Dengue fever, caused by dengue viruses, is a major health problem in tropical and subtropical regions of the world. The purpose of this study is to evaluate the safety of and immune response to a 2-dose regimen of a new monovalent dengue virus vaccine. This study will test the dengue virus vaccine DEN1delta30 in healthy adults.

DETAILED DESCRIPTION:
Dengue viruses account for more than 50 million cases of dengue fever and one half million cases annually of dengue hemorrhagic fever/shock syndrome. Dengue virus infections can cause illness ranging from mild, self-limited febrile illness to life threatening diseases. The goal of dengue vaccine development is to induce a long-lived antibody response against all four dengue serotypes. The rDEN1delta30 vaccine is a live attenuated dengue virus vaccine that may be protective against dengue serotype 1 (DEN1). The purpose of this study is to evaluate the safety, reactogenicity, and immunogenicity of a 2-dose regimen of rDEN1delta30 dengue virus vaccine. The regimen will differ in when the second booster shot of the vaccine is given.

This study will last 162 days (about 23 weeks) for those participants in Cohort 1, and 222 days (about 32 weeks) for those in Cohort 2. Participants in Cohort 1 will be randomly assigned to receive rDEN1delta30 vaccine or placebo on Study Day 0 and Study Day 120. Participants in Cohort 2 will be randomly assigned to receive rDEN1delta30 vaccine or placebo on Study Day 0 and Study Day 180.

There will be a total of 25 visits for each cohort. For both cohorts, the first and second vaccination days will include a physical exam and blood and urine collection, vital signs measurements, and receipt of the vaccine. A 30 minute observation period will follow vaccination. Participants will take their temperature at home three times a day for the first 16 days and report it in a diary. At all other study visits, vital signs measurements, a physical exam, and blood and/or urine collection will occur. At selected study visits, participants will turn in their diary cards.

Some participants may be asked to join an optional skin biopsy substudy.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Available for the duration of the study (23 weeks for Cohort 1 and 32 weeks for Cohort 2)
* Willing to use acceptable forms of contraception for the duration of the study

Exclusion Criteria:

* Clinically significant neurologic, heart, lung, liver, rheumatologic, autoimmune, or kidney disease
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, may interfere with the study
* Significant laboratory abnormalities
* Medical, work, or family problems as a result of alcohol or illegal drug use within 12 months prior to study entry
* History of severe allergic reaction or anaphylaxis
* Severe asthma
* HIV-1 infected
* Hepatitis C virus (HCV) infected
* Hepatitis B surface antigen positive
* Known immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive medications within 30 days prior to study entry. Individuals using topical or nasal corticosteroids are not excluded.
* Previous receipt of a live vaccine within 4 weeks prior to study entry
* Previous receipt of a killed vaccine within 2 weeks prior to study entry
* Absence of spleen
* Previous receipt of blood products within 6 months prior to study entry
* Previous receipt of dengue virus or other flavivirus (e.g., yellow fever virus, St.Louis encephalitis, West Nile virus) infection
* Previous receipt of yellow fever or dengue vaccine
* Plans to travel to an area where dengue infection is common
* Previous receipt of any investigational agent within 30 days prior to study entry
* Other condition that, in the opinion of the investigator, would affect participation in the study
* Pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To determine the safety and immunogenicity of a two-dose regimen of the rDEN1delta30 vaccine given as two doses separated by four or six months | Throughout study
To determine the optimum interval between first and second dose of rDEN1delta30 vaccine, as assessed by neutralizing antibody response to DEN1 induced by the vaccine | At 4 and 6 weeks after first and second vaccination

SECONDARY OUTCOMES:
To assess the frequency, quantity, and duration of viremia following each vaccine dose, based on the mean peak viremia, mean day of onset, and mean duration of viremia | Throughout study
To determine the number of vaccinees infected with rDEN1delta30 virus | Throughout study
To compare the infectivity rates, safety, and immunogenicity between dose 1 and 2 within a cohort and between cohorts | Throughout study
To evaluate the immunopathological mechanism of vaccine-associated rash in participants willing to undergo skin biopsy | Throughout study
To evaluate the phenotype and activation of peripheral blood mononuclear cells (PBMCs) at primary infection and challenge with DEN1 | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins School of Public Health
Locations (1):
- Center for Immunization Research, Johns Hopkins School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Blaney JE Jr, Sathe NS, Hanson CT, Firestone CY, Murphy BR, Whitehead SS. Vaccine candidates for dengue virus type 1 (DEN1) generated by replacement of the structural genes of rDEN4 and rDEN4Delta30 with those of DEN1. Virol J. 2007 Feb 28;4:23. doi: 10.1186/1743-422X-4-23. PMID 17328799
- [Background] Chaturvedi UC, Shrivastava R, Nagar R. Dengue vaccines: problems and prospects. Indian J Med Res. 2005 May;121(5):639-52. PMID 15937367
- [Background] Durbin AP, McArthur J, Marron JA, Blaney JE Jr, Thumar B, Wanionek K, Murphy BR, Whitehead SS. The live attenuated dengue serotype 1 vaccine rDEN1Delta30 is safe and highly immunogenic in healthy adult volunteers. Hum Vaccin. 2006 Jul-Aug;2(4):167-73. doi: 10.4161/hv.2.4.2944. Epub 2006 Jul 24. PMID 17012875
- [Background] Jacobs M, Young P. Dengue vaccines: preparing to roll back dengue. Curr Opin Investig Drugs. 2003 Feb;4(2):168-71. PMID 12669377
- [Background] Pang T. Vaccines for the prevention of neglected diseases--dengue fever. Curr Opin Biotechnol. 2003 Jun;14(3):332-6. doi: 10.1016/s0958-1669(03)00061-2. PMID 12849789
- [Background] Rothman AL. Dengue: defining protective versus pathologic immunity. J Clin Invest. 2004 Apr;113(7):946-51. doi: 10.1172/JCI21512. PMID 15057297
- [Background] Senanayake S. Dengue fever and dengue haemorrhagic fever--a diagnostic challenge. Aust Fam Physician. 2006 Aug;35(8):609-12. PMID 16894436
- [Derived] Katzelnick LC, Fonville JM, Gromowski GD, Bustos Arriaga J, Green A, James SL, Lau L, Montoya M, Wang C, VanBlargan LA, Russell CA, Thu HM, Pierson TC, Buchy P, Aaskov JG, Munoz-Jordan JL, Vasilakis N, Gibbons RV, Tesh RB, Osterhaus AD, Fouchier RA, Durbin A, Simmons CP, Holmes EC, Harris E, Whitehead SS, Smith DJ. Dengue viruses cluster antigenically but not as discrete serotypes. Science. 2015 Sep 18;349(6254):1338-43. doi: 10.1126/science.aac5017. PMID 26383952